CLINICAL TRIAL: NCT05613998
Title: Global Postural Reeducation vs. Non-specific Therapeutic Exercise in the Treatment of Rotator Cuff Tendinopathies of the Shoulder
Brief Title: Physiotherapy Treatment of Shoulder Rotator Cuff Tendinopathies. Global Postural Reeducation or Aerobic Exercise?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, Javier Álvarez, Principal Investigator, Universidad Francisco de Vitoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RPGEI
Record Dates: First submitted 2022-10-30; First posted 2022-11-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Tendinosis
Keywords: Tendinopathy; Rotator Cuff; Global Postural Reeducation; Aerobic Exercice; Shoulder Pain; Quality of life
MeSH Terms: conditions — Rotator Cuff Injuries; Tendinopathy; Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1. Global Postural Reeducation (GPR) intervention (Experimental): Patients who will receive the Global Postural Reeducation (GPR) treatment protocol
  Interventions: Other: GPR Group
- Group 2. Non-specific Aerobic exercice intervention (Experimental): Patients who will receive the non-specific aerobic exercise treatment protocol
  Interventions: Other: Aerobic Exercice Group
- Group 3. No physiotherapy intervention (No Intervention): Patients who will not receive physiotherapy treatment

INTERVENTIONS:
Other: GPR Group — 6-week treatment using the Global Postural Reeducation (GPR) method. 1 weekly session (45 min) with "frog on the ground" and "sitting" postures + daily home self-postures (10 min)
  Arms: Group 1. Global Postural Reeducation (GPR) intervention
Other: Aerobic Exercice Group — 6-week nonspecific aerobic exercise treatment. Participants will take a daily walk (20 min)
  Arms: Group 2. Non-specific Aerobic exercice intervention

SUMMARY:
The goal of this clinical trial is to compare in participant population (patients with rotator cuff tendinopathy of the shoulder) the effect of a Global Postural Reeducation (GPR) program vs. a nonspecific therapeutic (aerobic) exercise program

DETAILED DESCRIPTION:
Participants who meet the inclusion criteria will be randomly distributed between group 1 "Global Postural Reeducation (GPR)", group 2 "exercise", or group 3 "no physical therapy intervention".

Group 1 participants will receive a physical therapy treatment using the GPR method for 6 weeks consisting of 1 weekly session lasting 40 min performing "frog on the ground" and "sitting" poses. Patients in this group will also perform self-postures at home daily for 10 minutes.

Group 2 participants perform training for 6 weeks using non-specific aerobic exercise consisting of a daily 20-minutes walk at a speed of 4-5 km/h.

Group 3 participants will not receive any physical therapy treatment and will serve as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain with duration of at least 3 months
* Positive painful arc test during abduction
* At least one positive of the following tests: Hawkins-Kennedy test, Neer's sig, empty can test, drop arm or lift-off test

Exclusion Criteria:

* Cervical radiculopathy
* Moderate or severe degenerative arthropathy
* Complete rotator cuff tear
* History of shoulder or neck surgery
* History of shoulder fractures or dislocation
* Frozen shoulder or adhesive capsulitis
* Previous interventions with steroid injections or physiotherapy 2 months before the start of the program

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Changes in pain and disability after the treatment program | Baseline, one week after the last sessio, 3 months and 6 months after the last session
  Shoulder Pain and Disability Index (SPADI). Minimum value=0. Maximun value=100
Changes in pain and disability after the treatment program | Baseline, one week after the last sessio, 3 months and 6 months after the last session
  The Disabilities of the Arm, Shoulder and Hand (Quick-DASH). Minimum value=0. Maximun value=100

SECONDARY OUTCOMES:
Changes in pain after the treatment program | Baseline, one week after the last sessio, 3 months and 6 months after the last session
  Numerical Pain Rating Scale (NPRS). Minimum value=0 (no pain). Maximun value=10 (the worst pain imaginable)
Changes in pressure pain sensitivity | Pre, Post inmediate, and follow-up at 3 and 6 months
  Pressure Pain Thresholds (PPH)
Changes in Quality of Life | Baseline, one week after the last session, 3 months and 6 months after the last session
  Short-Form 12 Health Status Questionnaire. The response options form Likert-type scales that evaluate intensity or frequency.
  Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.
Changes in Range of Motion | Baseline, one week after the last sessio, 3 months and 6 months after the last session
  Goniometer

OTHER OUTCOMES:
Changes in stifness (cervical plexus, radial nerve, supraespinatus and infraespinatus muscles) | Baseline, one week after the last sessio, 3 months and 6 months after the last session
  Ultrasound Shear-Wave elastography

CONTACTS AND LOCATIONS:
Overall Officials: Javier Alvarez-González, Principal Investigator — Francisco de Vitoria University, Madrid, Spain; Arturo Morales-Muñiz, PhD, Study Director — Autonomous University of Madrid, Madrid, Spain; Alfredo Bravo-Sánchez, PhD, Study Chair — Francisco de Vitoria University, Madrid, Spain
Locations (1):
- Francisco de Vitoria University, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication
Access Criteria: Mail to the IP describing the interest and the purpose for accessing the data

REFERENCES:
- [Background] van der Heijden GJ, van der Windt DA, de Winter AF. Physiotherapy for patients with soft tissue shoulder disorders: a systematic review of randomised clinical trials. BMJ. 1997 Jul 5;315(7099):25-30. doi: 10.1136/bmj.315.7099.25. PMID 9233322
- [Background] Marinko LN, Chacko JM, Dalton D, Chacko CC. The effectiveness of therapeutic exercise for painful shoulder conditions: a meta-analysis. J Shoulder Elbow Surg. 2011 Dec;20(8):1351-9. doi: 10.1016/j.jse.2011.05.013. Epub 2011 Sep 1. PMID 21889366
- [Background] Littlewood C, Ashton J, Chance-Larsen K, May S, Sturrock B. Exercise for rotator cuff tendinopathy: a systematic review. Physiotherapy. 2012 Jun;98(2):101-9. doi: 10.1016/j.physio.2011.08.002. Epub 2011 Oct 5. PMID 22507359
- [Background] Kosek E, Ekholm J. Modulation of pressure pain thresholds during and following isometric contraction. Pain. 1995 Jun;61(3):481-486. doi: 10.1016/0304-3959(94)00217-3. PMID 7478692
- [Background] Naugle KM, Fillingim RB, Riley JL 3rd. A meta-analytic review of the hypoalgesic effects of exercise. J Pain. 2012 Dec;13(12):1139-50. doi: 10.1016/j.jpain.2012.09.006. Epub 2012 Nov 8. PMID 23141188
- [Background] Amorim CS, Gracitelli ME, Marques AP, Alves VL. Effectiveness of global postural reeducation compared to segmental exercises on function, pain, and quality of life of patients with scapular dyskinesis associated with neck pain: a preliminary clinical trial. J Manipulative Physiol Ther. 2014 Jul-Aug;37(6):441-7. doi: 10.1016/j.jmpt.2013.08.011. Epub 2014 Aug 3. PMID 25092553
- [Background] Heron SR, Woby SR, Thompson DP. Comparison of three types of exercise in the treatment of rotator cuff tendinopathy/shoulder impingement syndrome: A randomized controlled trial. Physiotherapy. 2017 Jun;103(2):167-173. doi: 10.1016/j.physio.2016.09.001. Epub 2016 Sep 21. PMID 27884499
- [Background] Kinsella R, Cowan SM, Watson L, Pizzari T. A comparison of isometric, isotonic concentric and isotonic eccentric exercises in the physiotherapy management of subacromial pain syndrome/rotator cuff tendinopathy: study protocol for a pilot randomised controlled trial. Pilot Feasibility Stud. 2017 Nov 14;3:45. doi: 10.1186/s40814-017-0190-3. eCollection 2017. PMID 29163981